CLINICAL TRIAL: NCT05655754
Title: A Prospective Randomized, Double Blind, Controlled, Safety and Non-inferiority Study of Esketamine Plus Propofol Compared to Methohexital Anesthesia for Electroconvulsive Therapy
Brief Title: Comparison of Esketamine/Propofol and Methohexital Anesthesia for ECT
Acronym: Ketofol
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Pia Baldinger-Melich, Assoc.Prof., Medical University of Vienna
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BMF22114
Record Dates: First submitted 2022-12-06; First posted 2022-12-19 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: ECT; Depression
Keywords: electroconvulsive therapy; depression; esketamine; anesthesia
MeSH Terms: conditions — Depression | interventions — Methohexital

STUDY DESIGN:
Intervention Model Description: Depressive patients, that are eligible for ECT, will be randomized to receiving either ECT with esketamine plus propofol or methohexital anesthesia for the whole series (min. 8 treatments). Participants and treating psychiatrists will be unaware or the anesthetic used; anesthetists will know the substance that it aministered during ECT. Both drugs will be compared in terms of safety, recovery time and clinical outcome.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Randomization of the study drug will be done using the software www.meduniwien.ac.at/randomizer according to consecutive CRF numbers. Stratification according to baseline HAMD17 scores (3 groups: HAMD 23-30, HAMD 30-40, HAMD>40), age and previous ECT (yes/no) will be performed Participants and treating psychiatrists will be unaware or the anesthetic used; anesthetists will know the substance that it aministered during ECT
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Methohexital (Active Comparator): Initial dose: methohexital 1 mg/kg (≙ 80 mg methohexital in a subject with 80 kg). If sufficient hypnosis is not achieved with the initial dose further doses of 10 mg methohexital will be administered until sufficient depth of anesthesia according to defined criteria is achieved. Criteria for sufficient depth of anesthesia will be comprised by a) the abolition of the eye-lash reflex b) absence of motor reaction upon inflation of the tourniquet.
  Maintenance dose: none (The drug combination is injected in order to initiate anesthesia) Route of administration: intravenous Duration: few seconds to initiate anesthesia. The procedure will be repeated for each ECT session.
  Interventions: Drug: Methohexital
- Ketofol (Active Comparator): Esketamine and propofol will be prepared shortly before injection by the nurse anesthetist as follows: 4 ml esketamine 25mg/ml, 6ml NaCl (0,9%), 10ml propofol (10mg/ml). The stability of ketamine-propofol mixtures (undiluted, 50:50 ratio) in one syringe has been documented for up to 3 hours.
  Initial dose: esketamine 0,5 mg/kg + propofol 0,5 mg/kg (≙ 40 mg esketamine + 40 mg propofol in a subject with 80 kg). If sufficient hypnosis is not achieved with the initial dose further doses of 5mg esketamine and 5 mg propofol will be administered until a sufficient depth of anesthesia is achieved.
  Maintenance dose: none (The drug combination is injected in order to initiate anesthesia) Route of administration: intravenous Duration: few seconds to initiate anesthesia. The procedure will be repeated for each ECT session
  Interventions: Drug: Ketofol

INTERVENTIONS:
Drug: Methohexital — anesthesia during ECT
  Arms: Methohexital
Drug: Ketofol — anesthesia during ECT
  Arms: Ketofol

SUMMARY:
The current anesthetic drug used as standard for ECT procedure at the Department of Psychiatry and Psychotherapy, Medical University of Vienna, is the barbiturate methohexital (Brevital®). As far as we know, methohexital is the most common anesthetic in the procedure of ECT. Only few heterogeneous randomized controlled trials to directly compare the use of (sole) ketamine and methohexital in ECT with relatively small sample sizes have been conducted so far, showing inconclusive findings: a retrospective comparison of methohexital and switch to ketamine anesthesia in 36 patients showed that ketamine prolonged seizure duration and accelerated posttreatment orientation. Others compared both drugs in terms of recovery and reorientation time showing that reorientation time was faster in the methohexital group (total N=9). Another study showed no difference in any outcome measure (depressive symptom improvement, cognition, adverse events) between both groups (total N=16, N=9 per group). Finally, a comparative investigation (total N=37, N=20 vs. N=17) detected no differences between both anesthetics but a higher systolic blood pressure posttreatment and longer motor seizure duration in the ketamine group. A favorable profile of ketamine in regards to seizure quality has been reported, however in terms of outcome measures methohexital and ketamine were similar (total N=50, N=23 vs. N=27).

The present study is designed as a prospective randomized non-inferiority trial comparing esketamine plus propofol (ratio 1:1, for better readability from now on referred to as "ketofol") to methohexital, the latter being the current standard anesthetic applied for ECT procedure at our department. Patients eligible for ECT will be randomly assigned to receive anesthesia with either ketofol or methohexital for the whole course of the individual ECT series. Group differences will be investigated both in regards to outcomes related to anesthesia, treatment-outcome and seizure quality.

Further, changes in cardiac enzyme levels before and after ECT-treatment and during the entire ECT series will be evaluated and possible group differences will be explored.

As stated above the sole/adjunct administration of ketamine as anesthetic agent for ECT has been associated with better seizure quality, similar antidepressant outcomes and anesthesia-associated events, while there is some evidence suggesting that the use of ketamine might present some advantages to other anesthetics in terms of cognitive side-effects accompanying ECT. Therefore, the aim of the present study will be to establish ketofol as a new standard for anesthesia at our Department.

ELIGIBILITY:
Inclusion Criteria:

* male or female inpatients
* age ≥ 18 years
* ICD-11 diagnosis of severe uni- or bipolar depression (F32.2, F32.2, F33.2, F33.3, F31.4, F31.5)
* Hamilton Depression Rating Scale HAMD17 ≥ 24
* ability to understand and willingness to sign written informed consent document
* negative urine pregnancy test in women
* anesthesiological approval for ECT (Classification of the American Society of Anesthesiologists ASA ≤ 3)
* antidepressant and antipsychotic medication in steady state for at least 7 days prior to first ECT treatment

Exclusion Criteria:

* severe somatic or neurological disease (esp. current or previous history of intracranial hypertension, uncontrolled severe hypertension, bleeds or aneurysm, recent myocardial infarction)
* current or past history of schizophrenia or schizoaffective disorder
* clinical relevant abnormalities on a general physical examination and routine laboratory screening
* pregnancy, breast feeding
* known allergy to the study drugs or compounds of the latter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
antidepressant effect | 4 weeks
  • HAMD17 change between baseline and post-ECT in both treatment arms over a series of 8 ECT sessions
recovery time | 4 weeks
  Mean recovery time over 8 ECT sessions in both treatment arms

SECONDARY OUTCOMES:
adverse events | 4 weeks
  AEs during anesthesia/ECT
concomitant medication | 4 weeks
  use of concom. medication during intervention to treat AEs
cognition | 4 weeks
  MMSE, Beck's Depression Inventory (BDI), multiple-choice word test (MWT-B), trail making test (TMT), reaction test (RT), cognitrone (COG), non-verbal learning test (NVLT), verbal learning test (VLT) (Vienna testing system, https://vts.schuhfried.com), compare cognitive outcomes before and after ECT in both treatment arms
time to reorientation | 4 weeks
  compare time to reorientation in both treatment arms
seizure quality | 4 weeks
  compare a function of seizure duration, concordance (seizure duration in the electromyogram/seizure duration in the electroencephalogram), midictal amplitude, peak heart rates and interhemispheric coherence in both treatment arms

CONTACTS AND LOCATIONS:
Locations (1):
- Pia Baldinger-Melich, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No